CLINICAL TRIAL: NCT03896204
Title: Effect of Telephone-supported Joint Protection Technique Training on Pain and Functionality in Lateral Epicondylitis
Brief Title: Effect of Telephone-supported Joint Protection Technique Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Özgü İnal, Assoc Prof, Trakya University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2019/32
Record Dates: First submitted 2019-03-28; First posted 2019-03-29 (Actual); Last update posted 2020-04-13 (Actual); Status verified 2020-04

CONDITIONS: Woman; Epicondylitis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- telephone-supported group (Experimental)
  Interventions: Behavioral: telephone-suppoted joint protection technique
- Other group (Experimental)
  Interventions: Behavioral: joint protection technique training

INTERVENTIONS:
Behavioral: telephone-suppoted joint protection technique — After joint protection technics training, patients will be followed up with telephone support for 1 month.
  Arms: telephone-supported group
Behavioral: joint protection technique training — Training will be given to individuals about joint protection technique
  Arms: Other group

SUMMARY:
There is limited evidence of the efficacy of joint protection principles in individuals diagnosed with lateral epicondylitis in the literature. The aim of this study was to investigate the effect of training of the telephone supported joint protection technique education on pain and upper extremity function in individuals with lateral epicondylitis. New information will be obtained according to the results.

DETAILED DESCRIPTION:
There is limited evidence of the efficacy of joint protection principles in individuals diagnosed with lateral epicondylitis in the literature. The aim of this study was to investigate the effect of training of the telephone supported joint protection technique education on pain and upper extremity function in individuals with lateral epicondylitis. New information will be obtained according to the results.

ELIGIBILITY:
* unilateral lateral epicondylitis diagnosis
* Individuals between 18-40

Exclusion Criteria:

-individuals with a history of surgery

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2019-03-29 (Actual); Primary Completion 2019-04-29 (Actual); Study Completion 2019-05-29 (Actual)

PRIMARY OUTCOMES:
hand grip strength | first month
  Jamar hand dynamometer; which has high validity and reliability across several studies and is therefore accepted as the gold standard for the measurement of hand grip strength.
pain and function | first month
  The Lateral Epicondylitis Function Scale; This scale is specially designed to evaluate patients with LE
function | first month
  The Upper Extremity Functional Index; Lower scores indicate increased difficulty with the relevant activity resulting from the subject's condition involving the upper limb
beahviour | first month
  Joint Protection Behavior Assessment-Short Form; evaluate the behavior of individuals during daily activities that require using the hands

CONTACTS AND LOCATIONS:
Overall Officials: Özgü İnal, Principal Investigator — Trakya University
Locations (1):
- Özgü İnal, Edirne, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided